CLINICAL TRIAL: NCT03215758
Title: A 12-week, Multicenter, Randomized, Double-blind, Placebo-controlled Study to Assess the Efficacy and Safety of QAW039 When Added to Standard-of-care Asthma Therapy in Patients With Uncontrolled Asthma
Brief Title: Study of Efficacy and Safety of QAW039 When Added to Standard-of-care Asthma Therapy in Patients With Uncontrolled Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CQAW039A2316; 2017-001273-16 (EudraCT Number)
Record Dates: First submitted 2017-07-11; First posted 2017-07-12 (Actual); Results first posted 2020-02-12 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: Asthma
Keywords: QAW039, uncontrolled asthma
MeSH Terms: conditions — Asthma | interventions — fevipiprant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- QAW039 (Active Comparator): QAW039 once daily
  Interventions: Drug: QAW039
- Placebo (Placebo Comparator): Placebo once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: QAW039 — QAW039 once daily
  Arms: QAW039
Drug: Placebo — Placebo once daily
  Arms: Placebo

SUMMARY:
A randomized, multicenter, double-blind, placebo- controlled parallel-group study to determine the efficacy and safety of QAW039, compared with placebo, when added to standard-of-care (SoC) asthma therapy in adult and adolescent (≥ 12 years) patients with uncontrolled asthma with respect to change from baseline in forced expiratory volume in 1 second (FEV1) at the end of 12 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of asthma (according to GINA 2016) for a period of at least 6 months.
* Treated with medium dose inhaled corticosteroid (ICS), or high dose ICS, or low dose ICS plus long- acting beta agonist (LABA), or low dose ICS plus leukotriene receptor antagonist (LTRA), or medium dose ICS plus LABA for at least 3 months prior to Visit 1 and the doses have been stable for at least 4 weeks prior to Visit 1.
* FEV1 of ≤85% for patients aged ≥18 years. FEV1 of ≤90% for patients aged 12 to <18 years.
* Daytime asthma symptom score (0 to 6 scale) of ≥1 per day during 4 of the last 7 days of the placebo run- in period.
* Total daily SABA use ≥1 puff per day during 4 of the last 7 days of the placebo run-in period.
* Demonstrated reversible airway obstruction.
* Asthma control questionnaire (ACQ) score ≥ 1.5.

Exclusion Criteria:

* Use of other investigational drugs within 5 half-lives of enrollment, or within 30 days, whichever is longer.
* A resting QTcF (Fridericia) ≥450 msec (male) or

  ≥460 msec (female).
* Pregnant or nursing (lactating) women.
* Serious co-morbidities.
* Patients on >20 mg of simvastatin, > 40 mg of atorvastatin, >40 mg of pravastatin, or >2 mg of pitavastatin.

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 675 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-07-02 (Actual); Study Completion 2019-07-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (101):
- United States (41):
  - Novartis Investigative Site, Flagstaff, Arizona
  - Novartis Investigative Site, Phoenix, Arizona
  - Novartis Investigative Site, Huntington Beach, California
  - Novartis Investigative Site, Long Beach, California
  - Novartis Investigative Site, Los Angeles, California
  - Novartis Investigative Site, Mission Viejo, California
  - Novartis Investigative Site, Mountain View, California
  - Novartis Investigative Site, Orange, California
  - Novartis Investigative Site, Roseville, California
  - Novartis Investigative Site, Walnut Creek, California
  - Novartis Investigative Site, Denver, Colorado
  - Novartis Investigative Site, Tamarac, Florida
  - Novartis Investigative Site, Winter Park, Florida
  - Novartis Investigative Site, Albany, Georgia
  - Novartis Investigative Site, Dacula, Georgia
  - Novartis Investigative Site, Honolulu, Hawaii
  - Novartis Investigative Site, Lihue, Hawaii
  - Novartis Investigative Site, Overland Park, Kansas
  - Novartis Investigative Site, Louisville, Kentucky
  - Novartis Investigative Site, Columbia, Missouri
  - Novartis Investigative Site, Rolla, Missouri
  - Novartis Investigative Site, Missoula, Montana
  - Novartis Investigative Site, Bellevue, Nebraska
  - Novartis Investigative Site, La Vista, Nebraska
  - Novartis Investigative Site, Skillman, New Jersey
  - Novartis Investigative Site, Asheville, North Carolina
  - Novartis Investigative Site, Gastonia, North Carolina
  - Novartis Investigative Site, High Point, North Carolina
  - Novartis Investigative Site, Cincinnati, Ohio
  - Novartis Investigative Site, Edmond, Oklahoma
  - Novartis Investigative Site, Eugene, Oregon
  - Novartis Investigative Site, Medford, Oregon
  - Novartis Investigative Site, Portland, Oregon
  - Novartis Investigative Site, Rapid City, South Dakota
  - Novartis Investigative Site, Boerne, Texas
  - Novartis Investigative Site, Dallas, Texas
  - Novartis Investigative Site, El Paso, Texas
  - Novartis Investigative Site, Fort Worth, Texas
  - Novartis Investigative Site, McKinney, Texas
  - Novartis Investigative Site, Seattle, Washington
  - Novartis Investigative Site, Greenfield, Wisconsin
- Argentina (13):
  - Novartis Investigative Site, Berazategui, Buenos Aires
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, Lanús, Buenos Aires
  - Novartis Investigative Site, Mar del Plata, Buenos Aires
  - Novartis Investigative Site, Santa Rosa, La Pampa Province
  - Novartis Investigative Site, Buenos Aires, Nueve De Julio
  - Novartis Investigative Site, Santa Fe, Rosario
  - Novartis Investigative Site, Rosario, Santa Fe Province
  - Novartis Investigative Site, San Miguel de Tucumán, Tucumán Province
  - Novartis Investigative Site, Buenos Aires
  - Novartis Investigative Site, Córdoba
  - Novartis Investigative Site, Mendoza
  - Novartis Investigative Site, Salta
- Germany (14):
  - Novartis Investigative Site, Peine, Lower Saxony
  - Novartis Investigative Site, Cottbus, Saxony
  - Novartis Investigative Site, Aschaffenburg
  - Novartis Investigative Site, Bamberg
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Fürstenwalde
  - Novartis Investigative Site, Gauting
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Lübeck
  - Novartis Investigative Site, Prien A Chiemsee
  - Novartis Investigative Site, Rüdersdorf
  - Novartis Investigative Site, Schleswig
  - Novartis Investigative Site, Schwerin
  - Novartis Investigative Site, Witten
- Hungary (6):
  - Novartis Investigative Site, Budaörs, HUN
  - Novartis Investigative Site, Ajka
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Debrecen
  - Novartis Investigative Site, Gödöllő
  - Novartis Investigative Site, Szeged
- Mexico (2):
  - Novartis Investigative Site, Culiacán, Sinaloa
  - Novartis Investigative Site, Río de Janeiro
- Philippines (4):
  - Novartis Investigative Site, Lipa City, Batangas
  - Novartis Investigative Site, Quezon City, Manila
  - Novartis Investigative Site, Iloilo City
  - Novartis Investigative Site, Manila
- Saudi Arabia (2):
  - Novartis Investigative Site, Riyadh, SAU
  - Novartis Investigative Site, Jeddah
- Slovakia (7):
  - Novartis Investigative Site, Bardejov, Slovak Republic
  - Novartis Investigative Site, Kežmarok
  - Novartis Investigative Site, Michalovce
  - Novartis Investigative Site, Poprad
  - Novartis Investigative Site, Prešov
  - Novartis Investigative Site, Spišská Nová Ves
  - Novartis Investigative Site, Žilina
- South Africa (5):
  - Novartis Investigative Site, Tygerberg, Cape Town
  - Novartis Investigative Site, Cape Town
  - Novartis Investigative Site, Chatsworth
  - Novartis Investigative Site, Durban
  - Novartis Investigative Site, Pretoria
- Turkey (Türkiye) (7):
  - Novartis Investigative Site, Istanbul, TUR
  - Novartis Investigative Site, Adana
  - Novartis Investigative Site, Ankara
  - Novartis Investigative Site, Istanbul
  - Novartis Investigative Site, Mersin
  - Novartis Investigative Site, Talas / Kayseri
  - Novartis Investigative Site, Yenisehir/Izmir

REFERENCES:
- See also: A Plain Language Trial Summary is available on novartisclinicaltrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=593
- See also: A Pediatric Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/ppatientsummary/ppatientsummaries?periodicPatientSummaryId=452

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from centers in Argentina (20), Germany (12), Hungary (4), Mexico (2), Philippines (4), Slovakia (7), South Africa (5), Turkey (5), United States (29)
Period: Overall Study
Arm/Group | QAW039 | Placebo
Started | 339 | 336
Completed | 334 | 328
Not Completed | 5 | 8
Not completed — Technical Problems | 1 | 0
Not completed — Protocol deviation | 0 | 1
Not completed — Physician Decision | 0 | 1
Not completed — Death | 0 | 1
Not completed — Adverse Event | 1 | 2
Not completed — Subject/Guardian Decision | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | QAW039 | Placebo | Total
Number analyzed (Participants) | 339 | 336 | 675
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48.1 (15.15) | 47.7 (15.40) | 47.9 (15.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 217 | 216 | 433
  Male | 122 | 120 | 242
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 274 | 281 | 555
  Black | 18 | 12 | 30
  Asian | 39 | 34 | 73
  Native American | 1 | 0 | 1
  Pacific Islander | 2 | 0 | 2
  Unknown | 0 | 3 | 3
  Other | 5 | 6 | 11

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Pre-dose FEV1 at Week 12
Description: Forced Expiratory Volume in one second (FEV1) is calculated as the volume of air forcibly exhaled in one second as measured by a spirometer. Baseline is defined as the last available FEV1 measurement taken prior to the first dose of randomized study drug.
Time Frame: Week 12
Population: Full analysis set (FAS): all randomized patients who received at least one dose of study medication. Patients in the FAS were analyzed according to the treatment they were assigned to at randomization.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | QAW039 | Placebo
Number analyzed (Participants) | 339 | 336
Liters | 0.112 (0.0167) | 0.071 (0.0169)
Statistical Analysis 1: Comparison: QAW039 vs Placebo; Test type: Superiority; p = 0.088, ANCOVA; Mean Difference (Net) = 0.0238, 95% CI 2-sided [-0.006 to 0.088]

2. Secondary Outcome: Change From Baseline in Daytime Asthma Symptom Score
Description: Daytime asthma symptoms are evaluated through four questions and each of them will be rated on a scale of 0 to 6. Higher scores indicate more severe asthma-related symptoms. A mean score will be calculated for the responses to 4 questions.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score
Arm/Group | QAW039 | Placebo
Number analyzed (Participants) | 339 | 336
Score | -0.56 (0.036) | -0.51 (0.037)
Statistical Analysis 1: Comparison: QAW039 vs Placebo; Test type: Superiority; p = 0.278, ANCOVA; Mean Difference (Net) = -0.06, 95% CI 2-sided [-0.16 to 0.05]

3. Secondary Outcome: Change From Baseline in Daily Use of SABA
Description: Daily use of SABA (the number of rescue medication puffs taken in the previous 12 hours) was recorded using a patient electronic diary (referred to as eDiary or eDiary/ePEF). Patients were instructed to routinely complete the patient diary twice daily - at the same time each morning and each evening, approximately 12 hours apart.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Number of puffs
Arm/Group | QAW039 | Placebo
Number analyzed (Participants) | 339 | 336
Number of puffs | -1.11 (0.075) | -1.02 (0.076)
Statistical Analysis 1: Comparison: QAW039 vs Placebo; Test type: Superiority; p = 0.429, ANCOVA; Mean Difference (Net) = -0.08, 95% CI 2-sided [-0.30 to 0.13]

4. Secondary Outcome: Change From Baseline in Asthma Quality of Life (AQLQ+12) Score
Description: AQLQ is a 32-item instrument administered as a self-assessment. AQLQ+12 is a modified version of AQLQ developed to measure functional impairments of participants aged 12-70 years. It is divided into 4 domains: activity limitation, symptoms, emotional function, and environmental stimuli. Participants were asked to recall their experiences during the last 2 weeks and respond to each question on a 7-point scale (1=severe impairment, 7=no impairment), where higher scores indicated "better quality of life." Overall AQLQ+12 score is the mean of all 32 responses.
Time Frame: Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | QAW039 | Placebo
Number analyzed (Participants) | 339 | 336
units on a scale | 0.91 (0.048) | 0.89 (0.049)
Statistical Analysis 1: Comparison: QAW039 vs Placebo; Test type: Superiority; p = 0.777, ANCOVA; Mean Difference (Net) = 0.069, 95% CI 2-sided [-0.12 to 0.15]

ADVERSE EVENTS:
Time Frame: After signing informed consent to 30 days after last dose
Groups:
- QAW039 150 mg: QAW039 150 mg
- Placebo: Placebo
Arm/Group | QAW039 150 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/339 | 1/336
Serious Adverse Events (participants affected / at risk) | 1/339 | 5/336
Other Adverse Events (participants affected / at risk) | 94/339 | 102/336
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | QAW039 150 mg (N=339) | Placebo (N=336)
Upper respiratory tract infection bacterial (Infections and infestations) | 0 | 1
Electrocardiogram T wave inversion (Investigations) | 0 | 1
Astrocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | QAW039 150 mg (N=339) | Placebo (N=336)
Diarrhoea (Gastrointestinal disorders) | 2 | 4
Fatigue (General disorders) | 2 | 4
Acute sinusitis (Infections and infestations) | 4 | 1
Bronchitis (Infections and infestations) | 12 | 10
Nasopharyngitis (Infections and infestations) | 13 | 12
Rhinitis (Infections and infestations) | 1 | 5
Upper respiratory tract infection (Infections and infestations) | 6 | 10
Upper respiratory tract infection bacterial (Infections and infestations) | 5 | 5
Viral upper respiratory tract infection (Infections and infestations) | 7 | 6
Blood creatine phosphokinase increased (Investigations) | 2 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 4
Headache (Nervous system disorders) | 6 | 7
Asthma (Respiratory, thoracic and mediastinal disorders) | 43 | 45
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 5
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 12 | 6
Hypertension (Vascular disorders) | 1 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-05-10): https://cdn.clinicaltrials.gov/large-docs/58/NCT03215758/Prot_001.pdf
  • Statistical Analysis Plan (2019-08-25): https://cdn.clinicaltrials.gov/large-docs/58/NCT03215758/SAP_000.pdf